CLINICAL TRIAL: NCT05803148
Title: Effect of Cardioneuroablation vs Midodrine on Syncope Recurrence Among Patients With Vasovagal Syncope: The CAMPAIGN Randomized Clinical Trial
Brief Title: Treatment Strategy of Vasovagal Syncope
Acronym: CAMPAIGN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Beijing Chao Yang Hospital (Other); RenJi Hospital (Other); Yeditepe University Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Ningbo No. 1 Hospital (Other); Fuwai Yunnan Cardiovascular Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yan Yao, MD,PhD, Chief of First Department of Arrythmia Center, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-GSP-QZ-4
Record Dates: First submitted 2023-03-09; First posted 2023-04-07 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Syncope, Vasovagal
Keywords: Vasovagal syncope; Cardioneuroablation; Midodrine
MeSH Terms: conditions — Syncope, Vasovagal | interventions — Midodrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Cardioneuroablation (Experimental): In this arm, the catheter ablation of the GPs will be performed in the order of LSGP, LIGP, RIGP, left atrial RAGP and right atrial RAGP. Patient education includes fully informing patients of the benign prognosis of vasovagal syncope, and educating patients to avoid triggering factors as much as possible. At the same time, the patient should be taught how to cope with the impending syncope with physical counter-pressure maneuvers and dietary suggestions that emphasize fluid and sodium intake.
  Interventions: Procedure: Cardioneuroablation
- Control group: Midodrine (Active Comparator): In this arm, Midodrine will be applied without the following contraindications: hypertension, chromaffin cell carcinoma, acute nephritis, severe renal dysfunction, glaucoma, prostatic hyperplasia with urinary retention, mechanical urinary obstruction, hyperthyroidism. Patient education includes fully informing patients of the benign prognosis of vasovagal syncope, and educating patients to avoid triggering factors as much as possible. At the same time, the patient should be taught how to cope with the impending syncope with physical counter-pressure maneuvers and dietary suggestions that emphasize fluid and sodium intake.
  Interventions: Drug: Midodrine Oral Tablet

INTERVENTIONS:
Procedure: Cardioneuroablation — The left atrium model was established under the guidance of three-dimensional mapping. Atrial septum puncture、left atrium mapping and right atrium mapping will be performed according to standard EP lab protocol. The location of GPs will be detected with HAFE potential (duration ≥ 50ms， deflections ≥ 4 times， amplitude ≥ 0.7mV) and high frequency stimulation (HFS; 30 Hz, 20 mV, pulse width 2ms) through positive vasovagal response (transient ventricular asystole, atrioventricular block, or R-R interval increased by 30%) . Saline Irrigated-tip catheter with pressure monitoring will be applied for the procedure, and radiofrequency energy is limited to 40W and 43℃ for at least 30s at each site. The ablation endpoint for each GP is defined as the complete elimination of all targeted HAFE potential and elimination of positive vasovagal response. The endpoint of the procedure was that the heart rate reach 75% of the maximum heart rate in atropine test.
  Other Names: Cardiac ganglion plexus ablation
  Arms: Experimental group: Cardioneuroablation
Drug: Midodrine Oral Tablet — Midodrine will start dosing with 5 mg of the study drug 3 times daily, 4 hours apart, during daylight hours.Dose with be adjusted within a range of 2.5 mg twice daily, 4 hours apart, up to 10 mg, 3 times daily, every 4 hours. The optimal dose ranging be completed within the first 2 weeks. If intolerable symptoms persisted despite dose reductions, the drug will be withdrawn, and the patient was released from the study.
  Other Names: Midodrine pill
  Arms: Control group: Midodrine

SUMMARY:
This is a prospective, international multi-center, open-labeled, randomized trial.

The investigator speculated that CNA prevents more patients with moderate to severe VVS from syncope recurrence compared to midodrine.

DETAILED DESCRIPTION:
Nearly 40% of people faint at least once in their life, and vasovagal syncope (VVS) is the most common cause. Study shows that VVS accounts for 66% of syncope in the Emergency Room. The early peak incidence is around 15 years for young women and a later significant rise in visits for both sexes over the age of 65 years. Patients with frequent syncope have a markedly reduced quality of life, similar to that of patients with severe rheumatoid arthritis or chronic low back pain.

Vasovagal syncope is characterized by paroxysmal hypotension and/or bradycardia. Multiple hypotheses have been suggested as the mechanism of VVS, hence the treatment was diverse. The current therapy suggested by guidelines includes diet, counter-pressure maneuvers, beta-blockers, fludrocortisone, serotonin reuptake inhibitors, midodrine, and permanent pacemakers.

Cardioneuroablation (CNA) which modified the cardiac autonomic nervous system through catheter ablation shows encouraging results in preventing syncope recurrence. Experience from our center also suggested that CNA was highly effective, with a syncope-free rate of nearly 80% for 4-year follow-up; however, the studies were non-randomized with no control group. A recent single-center randomized control study has reported that CNA was superior to non-pharmacology therapy for syncope prevention. The investigators are hereby willing to compare the effectiveness of CNA to drug therapy in a multi-center randomized control fashion.

The objective of this trial is to determine the role of CNA and midodrine therapy in the prevention of syncope recurrence in patients with vasovagal syncope and provide evidence for clinical treatment strategies. Participants will be randomized to either CNA plus patient education (diet, avoidance trigger, physical counter-pressure maneuvers) or midodrine therapy plus patient education. Randomization will be carried out with interactive web response system stratified by center.

The participants were followed up at 7 days, 3 months, 6 months, 12 months and 24 months respectively after ablation procedure, to observe whether there were recurrent syncope and /or pre-syncope (including the time and frequency of recurrent syncope, inducing factors, and whether complicated with fall injury, etc.), and to reassessed tilt test, 24-hour ambulatory electrocardiogram and fill in Euroqol (EQ-5D) and ISQL quality of life score form. To evaluate the safety and efficacy of cardiac nerve ablation in the prevention of refractory vasovagal syncope. The tilt test, the changes of vagus nerve function and the improvement of quality of life before and after were analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age
2. Calgary Syncope Symptom Score ≥ -2 points
3. Positive response to head-up tilt test
4. With syncope episodes more than 3 times in the preceding year
5. A proven failure of non-pharmacologic treatment, including reassurance regarding the benign prognosis, education about the avoidance of situations and triggers initiating syncope， application of PCM during the occurrence of prodromal symptoms, and lifestyle modifications（adequate fluid intake and salt supplementation）， according to the guideline
6. Willingness to comply with follow-up requirements and to sign the informed consent

Exclusion Criteria:

1. Complied with other causes of syncope, including postural hypotension, aortic stenosis, sick sinus node syndrome, high-grade atrioventricular block, ventricular arrhythmias, pulmonary hypertension, hypertrophic cardiomyopathy, transient ischemic attack, epilepsy, sequelae of cerebral infarction or cerebral hemorrhage, subclavian vein steal syndrome and drug-induced syncope.
2. Complied with congenital heart disease, valvular heart disease, cardiomyopathy, and diabetes.
3. History of cardiac catheter ablation, peacemaker implantation and cardiac surgery.
4. History of midodrine usage, or compiled with contradiction of midodrine, including urine retention, hypertension (Bp≥140/90mmHg), glaucoma， renal dysfunction.
5. Life expectancy <1 year for any medical condition
6. Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with syncope recurrence during follow-up | 12 month after randomization
  Syncope was defined as a transient loss of consciousness and complete recovery in a very short time.

SECONDARY OUTCOMES:
Number of Participants with pre-syncope during follow-up | 12 month after randomization
  Pre-syncope was defined as the prodrome before syncope, such as dizziness, sweating，dyspnea, and paleness, and patients did not actually fall down. We documented each time that syncope occurred. The severeity of the prodrome will be assessed with a standardized questionnaire CPF.
Quality of life measure by Impact of Syncope on Quality of Life（ISQL）questionnaire | 6 month after randomization
  The difference in quality of life between the two groups as compared to baseline by using the standardized ISQL (Impact of Syncope on Quality of Life) questionnaire. The ISQL score was ranged from 0 to 57 points, and higher points represented more severe impaired quality of life.
Quality of life measure by Impact of Syncope on Quality of Life（ISQL）questionnaire | 12 month after randomization
  The difference in quality of life between the two groups as compared to baseline by using the standardized ISQL (Impact of Syncope on Quality of Life) questionnaire. The ISQL score was ranged from 0 to 57 points, and higher points represented more severe impaired quality of life.
Results of Head-up tilt test | 12 month after randomization
  The difference in the rate of head-up tilt test induced syncope between the two groups. The positive results of head-upright tilt test were defined by VASIS standard. The examination will be performed at each investigative center.
Blood pressure measured with 24 hours monitoring | 6 month after randomization
  The difference in blood pressure between the two groups as compared to baseline. Both systolic and diastolic blood pressure were assessed. The device provided to patients prior to discharge or at outpatient visits will be used for this assessment.
Blood pressure measured with 24 hours monitoring | 12 months after ablation procedure
  The difference in blood pressure between the two groups as compared to baseline. Both systolic and diastolic blood pressure were assessed. The device provided to patients prior to discharge or at outpatient visits will be used for this assessment.

CONTACTS AND LOCATIONS:
Overall Officials: yan Yao, PhD, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tu B, Wu L, Hu F, Fan S, Liu S, Liu L, Ding L, Zheng L, Yao Y. Cardiac deceleration capacity as an indicator for cardioneuroablation in patients with refractory vasovagal syncope. Heart Rhythm. 2022 Apr;19(4):562-569. doi: 10.1016/j.hrthm.2021.12.007. Epub 2021 Dec 9. PMID 34896621
- [Result] Sheldon R, Faris P, Tang A, Ayala-Paredes F, Guzman J, Marquez M, Morillo CA, Krahn AD, Kus T, Ritchie D, Safdar S, Maxey C, Raj SR; POST 4 investigators. Midodrine for the Prevention of Vasovagal Syncope : A Randomized Clinical Trial. Ann Intern Med. 2021 Oct;174(10):1349-1356. doi: 10.7326/M20-5415. Epub 2021 Aug 3. PMID 34339231
- [Result] Hu F, Zheng L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Right anterior ganglionated plexus: The primary target of cardioneuroablation? Heart Rhythm. 2019 Oct;16(10):1545-1551. doi: 10.1016/j.hrthm.2019.07.018. Epub 2019 Jul 19. PMID 31330187
- [Derived] Maimaitijiang P, Tu B, Lai Z, Chen A, Zhang Z, Zhou L, Cai S, Zheng L, Yao Y; CAMPAIGN Investigators. The Efficacy of Cardioneuroablation versus Midodrine in Patients with Vasovagal Syncope: Design and Rationale for the CAMPAIGN Trial. J Interv Card Electrophysiol. 2025 Mar;68(2):257-265. doi: 10.1007/s10840-025-02029-4. Epub 2025 Mar 21. PMID 40117099